CLINICAL TRIAL: NCT02044107
Title: Measuring the Effectiveness of Co-packaging to Improve Provider and Caregiver Behavior in the Treatment of Diarrhea With Zinc & ORS and Pneumonia With Zinc & Antibiotics for Children Under 5 Yrs From San Marcos, Guatemala
Brief Title: The Effectiveness of Co-packaging With Zinc to Improve Treatment of Diarrhea and Pneumonia in Guatemala
Acronym: Zinc10
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Center for Studies of Sensory Impairment, Aging and Metabolism (Other)
Collaborators: Micronutrient Initiative (Other)
Responsible Party: Principal Investigator, Marieke Vossenaar, Senior Program Leader for Diet and Health, Center for Studies of Sensory Impairment, Aging and Metabolism
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CeSSIAM_01
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Diarrhea.; Pneumonia.
Keywords: Diarrhea,; Pneumonia,; Zinc treatment,; Patient Compliance.
MeSH Terms: conditions — Diarrhea; Pneumonia; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Co-packaging and counseling messages (Experimental): Current standard care at public health center ( zinc ORS for treatment of diarrhea and antibiotics for treatment of of pneumonia).
  The intervention consists of health center level co-packaging and visual counseling messages (zinc & ORS packaged at health center for diarrhea, and zinc & antibiotics co-packaged at health center for pneumonia) Co-packaging is done in a plastic bag, which is covered with pre-tested zinc treatment messages - a distinct packaging has been designed for diarrhea and for pneumonia
  Interventions: Behavioral: Co-packaging and counseling messages
- Control group (No Intervention): Current standard care at public health center (zinc & ORS for treatment of diarrhea and zinc & antibiotics for treatment of of pneumonia).

INTERVENTIONS:
Behavioral: Co-packaging and counseling messages — The intervention involves co-packaging in 2 distinct packages: 1) for diarrhea treatment to package zinc & ORS for the treatment of diarrhea using a plastic bag with printed messages that were pre-tested in formative research; and 2) for pneumonia treatment to co-package zinc & antibiotics in a plastic bag with printed messages that were pre-tested in a formative research phase. Pre-tested zinc treatment messages will be on posters displayed in the intervention health centers. Orientation will be provided to health facility staff in control and intervention areas.
  Other Names: The physical co-packaging is called the "bolsita salva-vida"
  Arms: Co-packaging and counseling messages

SUMMARY:
This project applies a randomized community design to test the effectiveness of health center level co-packaging and counseling messages to improve provider and caregiver behavior in the treatment of diarrhea with zinc & oral rehydration salts (ORS) and treatment of pneumonia with zinc & antibiotics in children aged 2-59 mo old. We will evaluate the adherence of caregivers in 10 health posts in 5 municipalities randomly assigned to receive the health center level co-packaging and counseling messages in addition to current standard care, by comparing them with the caregivers in 10 health posts in 5 municipalities randomly assigned to the receive only the current standard of care. Cost-effectiveness of co-packaging at the health-center level, as a means of improving provider treatment and counseling practices and caregiver adherence, will be evaluated.

The main objective is to establish the effectiveness of a facility level co-packaging and counseling messages for increasing the adherence by caregivers of children aged 2-59 mo old to the prescribed 10 day treatment with zinc to complement ORS for the treatment of diarrhea and zinc to complement the antibiotics for the treatment of pneumonia diagnosed and treated in public health posts.

Specific Quantitative Objectives:

• To determine if visible co-packaging with pre-tested counseling messages:

* Improves adherence of caregivers of children towards the prescribed zinc treatment.
* Improves knowledge, awareness or attitudes of caregivers of children and health providers at public health care centers towards the prescribed zinc treatment.
* Results in overall increase in health care-seeking for the treatment of diarrhea and pneumonia at public health care centers.

Specific Qualitative Objectives:

* To establish the perception, attitudes and experiences of caregivers towards the visible co-packaging with pre-tested counseling messages to promote the prescribed zinc treatment.
* To establish the perception, attitudes and experiences of health providers at public health care centers towards the visible co-packaging with pre-tested counseling messages to promote the prescribed zinc treatment.
* To establish the perception, attitudes and experiences of children aged 4 to 5 years old towards the visible co-packaging with pre-tested counseling messages to promote the prescribed zinc treatment.

DETAILED DESCRIPTION:
Please note that the study protocol is also available in Spanish.

ELIGIBILITY:
Inclusion Criteria:

* The child is aged between between 2 and 59 mo old (< 5 years old).
* The child is diagnosed with diarrhea or pneumonia at one of the selected public health care centers.
* The caregiver accompanying the child to the public health care centers must live in the same household.

Exclusion Criteria:

* Unwillingness to sign consent form.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of caregivers who administer zinc to child for at least 8 days. | 10 days
  Improved adherence to diarrhea or pneumonia treatment with zinc for the prescribed 10 days based on pill count in the home.
  Expressed as percentage of caregivers who administer zinc to child for at least 8 days.
Percentage of caregivers who report giving zinc to child for at least 8 days. | 10 days
  Improved adherence to diarrhea or pneumonia treatment with zinc for the prescribed 10 days based on self-reports.
  Expressed as percentage of caregivers who report administering zinc to child for at least 8 days.

SECONDARY OUTCOMES:
Improved Provision of Care for Treatment of Diarrhea and Pneumonia | 6 months
  Percentage of caregivers who receive zinc from the health post. Percentage of caregivers that reported receiving instructions on how to prepare zinc.
  Percentage of caregivers that report favorable experience with treatment from the health center.
  Percentage of caregivers that report favorable experience with packaging

CONTACTS AND LOCATIONS:
Overall Officials: Marion Roche, PhD, Study Director — Micronutrient Initiative; María del Rosario García Meza, MA, Principal Investigator — Center for Studies of Sensory Impairment, Aging and Metabolism; Noel W Solomons, MD, Study Chair — Center for Studies of Sensory Impairment, Aging and Metabolism; Marieke Vossenaar, PhD, Principal Investigator — Center for Studies of Sensory Impairment, Aging and Metabolism
Locations (1):
- Guatemala: Ministry of Public Health and Social Assistance, San Marcos, Departamento de San Marcos, Guatemala